CLINICAL TRIAL: NCT00618527
Title: Combination Therapy Using Mycophenolate Mofetil (CellCept) and Human Interferon beta1a (Rebif) in Early Treatment of Multiple Sclerosis
Brief Title: Combination Therapy Using Cellcept and Rebif in RRMS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aaron Boster (Other)
Collaborators: EMD Serono (Industry); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Aaron Boster, Assistant Professor-Clinical, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006H0039
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Multiple Sclerosis
Keywords: relapsing remitting multiple sclerosis; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Mycophenolic Acid; Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Rebif with Cellcept
  Interventions: Drug: mycophenolate mofetil (Cellcept); Drug: human interferon beta 1a (Rebif)
- 2 (Placebo Comparator): Rebif alone
  Interventions: Drug: human interferon beta 1a (Rebif)

INTERVENTIONS:
Drug: mycophenolate mofetil (Cellcept) — 1 gram po, bid
  Other Names: Cellcept
  Arms: 1
Drug: human interferon beta 1a (Rebif) — 44mcg sq injection every other day
  Other Names: Rebif

SUMMARY:
The purpose of this trial is to examine the benefits of early combination of CellCept® with Rebif® in long-term management of patients with multiple sclerosis. Quantitation of mRNA for MxA gene from ex-vivo lymphocytes obtained from patients receiving both drugs or interferon alone will be used to gauge the usefulness of this combination therapy. In addition we will examine the safety of combination of mycophenolate mofetil and interferon beta 1a in treatment of multiple sclerosis.

This is a pilot study to examine if the combination of CellCept® with Rebif® will prove to be useful in the early treatment of patients with MS. Up-regulation of the MxA gene following the administration of Rebif® will be used as a surrogate marker of interferon bioactivity. This in turn could serve as a surrogate marker of interferon efficacy in these patients.

The null hypothesis is that there will not be any difference in the proportion of patients that produce MxA gene transcripts in the Rebif® group as compared to the group that received Rebif® with CellCept® at the end of this study (1 year).

The alternate hypothesis is that the combination of CellCept® with Rebif® will prove to be useful in prolonging the efficacy of interferon. In other words, the combination will result in a significant proportion of patients in the treatment group continuing to produce MxA as compared to the proportion of patients producing MxA in the Rebif® arm.

DETAILED DESCRIPTION:
A total of 30 patients will be studied, fifteen in each arm. Proportional analysis for sample size estimation could not be done since the proportion of MxA positive patients at 1 year in the Rebif® treatment arm is unknown. Nevertheless, a sample size of 15 patients per arm will allow the detection of a suitable difference between the treatment groups as outlined below:

For purposes of this study an MxA non-producer will be designated as a "treatment failure" irrespective of the clinical status. The definition of an MxA non-producer is a patient who is producing 1 year into treatment; MxA transcripts at a level 2 SD below his/her mean baseline value at entry. Accordingly, patients will be compared to their own initial response to Rebif® at entry into the study. In the following examples the proportion of MxA non-producers in each group will be used for comparisons.

At the end of 1 year, the incidence of neutralizing antibodies in patients receiving Rebif® 44 micrograms SC tiw is approximately 20%. For purposes of calculation of sample size, a proportion of 40% (0.4) was chosen for the MxA non-producers in the Rebif® arm, since the proportion of patients that fail to produce MxA at 1 year is higher than the proportion that show neutralizing antibodies. In other words, mechanisms other than neutralizing antibodies are the basis of interferon unresponsiveness in most patients, an important phenomenon that is lost to detection if the sole focus is restricted to neutralizing antibodies. Assuming that the combination will be effective in maintaining biological activity of interferon at 1 year in most or all of the patients, the following scenarios can be identified.

Patients will be randomly assigned to either receive Rebif with or without CellCept. The randomization process will utilize a computer program designed specifically for randomizing patients. Patients will have an equal chance of being randomized to receive Rebif with or without CellCept therapy.

Each subject must meet the following eligibility criteria (i.e., all of the Inclusion criteria and not of the Exclusion criteria) before enrollment in to the study:

Inclusion Criteria

* Male and female subjects clinically eligible for interferon therapy, including a diagnosis of relapsing multiple sclerosis (according to the MacDonald criteria, revised 2005), or patients diagnosed with clinically isolated syndrome.
* Patients must be between the ages of 18 to 65, inclusive
* Subjects must have adequate cognitive function to understand and sign the IRB-approved consent prior to the performance of any study-specific procedures.

Exclusion Criteria

* Females who are pregnant or breastfeeding, and females of childbearing potential (i.e. not surgically sterile or at least two years postmenopausal) who engage in active heterosexual relations, and have not had a hysterectomy or bilateral oophorectomy, and are not using one of the following birth control methods: tubal ligation, implantable contraceptive device, oral, patch or injectable contraceptive, barrier method, or sexual activity restricted to vasectomized partner will be excluded from this study due to the potential risk to the unborn fetus and/or nursing infant.
* Subject has clinically significant abnormal laboratory values. An abnormal value is defined as CTCAE Version 3.0, Grade 2 or worse lab value determined to be clinically significant by the Principal Investigator.
* Subject has received corticosteroids within 30 days prior to the screening visit.
* Subject has received cyclophosphamide or mitoxantrone.
* Subject has received Imuran or methotrexate in the last 3 months.
* Subject has any medical condition, or history of a medical condition, that would interfere with the interpretation of the study results or the conduct of the study as determined by the investigator. This may include other autoimmune disease, history of cancer, uncontrolled hypertension, myelodysplastic syndromes and any other uncontrolled cardiac, hepatic, renal or pulmonary history as determined by the investigator to be clinically significant.
* Subject is participating or has participated in another clinical trial or received another investigational therapy in the last 90 days.

Primary measures of efficacy:

* Analysis of the proportion of patients who are MxA producers in the group receiving Rebif® with CellCept®, as compared to the proportion of patients on Rebif® alone who are MxA producers.
* Comparison of the mean MxA levels in the Rebif® with CellCept® group to that of Rebif® alone.

The null hypothesis is that there will not be any difference between the two treatment arms regarding the levels of mRNA for MxA. The alternate hypothesis is that the treatment arm will have a sustained high level of mRNA as compared to the Rebif® alone treatment group.

Secondary measures of efficacy

* Clinical status, including number and severity of clinical exacerbations, severity of exacerbations, time to first and second exacerbations, disability as measured by Expanded Disability Status Scale (EDSS) and Multiple Sclerosis Functional Composite (MSFC) and use of corticosteroids during the 1 year study.
* Tolerance to interferon and clinical burden of disease as measured by the Multiple Sclerosis Quality of Life Index (MSQLI).
* Break-through disease as detected by gadolinium enhancement of lesions in MRI at the conclusion of the study.
* Total burden of T2 FLAIR disease in the combination arm as compared to Rebif® alone at the conclusion of the study.

Measuring MxA

MxA levels in patients will be determined by measuring relative amounts of MxA mRNA in peripheral blood mononuclear cells (PBMCs) isolated from their blood. Blood will be collected in preservative free heparin tubes and the PBMCs isolated by Ficoll-Histopaque gradient centrifugation. The PBMCs will be harvested, washed, and the total cell counts established. Total RNA will be isolated from these cells. RNA will then be converted to cDNA in a reverse transcription reaction.

Real-time polymerase chain reaction (PCR) will be performed to establish levels of gene activation of MxA. As in standard PCR, oligonucleotide primers and temperature cycling are used to amplify the target sequence from the template DNA. With real-time PCR, an oligonucleotide "probe" is added to the mix. This probe has a high-energy "reporter" dye at the 5' end and a low-energy "quencher" dye at the 3' end. The probe is designed to anneal to a specific portion of the target DNA sequence. When the probe is intact, the proximity of the quencher dye to the reporter dye suppresses its natural fluorescence. As DNA polymerase makes copies of the template DNA molecules in the mix, the attached probe is cleaved, and the distance between the reporter and quencher dyes increases, causing fluorescent emission by the reporter to also increase. Fluorescence is measured throughout the temperature cycles of the PCR reaction. Calculations are made based on the detected fluorescence to determine the amount of initial template DNA that was present in the sample. Because it is impossible to determine the exact number of MxA mRNA molecules that each sample started with, real-time PCR is done to detect levels of GAPDH, a standard housekeeping gene, in each sample so that a comparison between GAPDH and MxA can be made, and relative quantities can be determined between different samples.

Measuring T2 FLAIR Total burden of T2 FLAIR is measured by a semi-automated computer program used within the radiology department. The software will outline all lesions within the scanned area. Once mapped out, the MRIs will be reviewed by Dr. Eric Bourekas for measurement and quantification of total disease burden.

Detailed study procedures

Treatment Schedule Eligible patients will be randomized to receive treatment with or without mycophenolate mofetil 2,000 mg per day for 6 months. After 4 weeks of therapy both groups will receive Rebif® at the standard dose of 44 micrograms SC TIW, after a standard titration dosing regimen. Patients will be evaluated every 3 months for one year. The patient's total time on study will be one year.

Randomization will occur at the Day 0 visit and will utilize a computer program specifically created for this purpose. Patients will have a 50% chance of receiving CellCept.

End of Study

If a patient develops any medical condition that, in the opinion of the investigator, would make it unsafe for them to continue on the study, the patient will be removed from study and followed off study for safety, resolution of any event. Patient removal from study will be evaluated on a case by case basis at the investigators discretion and will be carried out to ensure the patients safety.

If a patient experiences greater than 2 exacerbations requiring corticosteroid therapy (moderate to severe) in any 12 month period, or have confirmed progression in Expanded Disability Status Scale (EDSS) of > 2 points with or without exacerbations they would be considered treatment failures for the appropriate treatment arm and would be removed from the study to pursue other treatment options.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with relapsing remitting multiple sclerosis
* eligible to initiate interferon therapy
* between he ages of 18-65, inclusive

Exclusion Criteria:

* have received corticosteroids within 30 days prior to study start
* have ever received cyclophosphamide or mitoxantrone
* have received Imuran or methotrexate in the last 3 months
* females that are pregnant or breastfeeding are excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
mRNA for MxA gene levels | Day 0, Week 4, Week 16, Week 28, Week 40, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Aaron L Boster, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Multiple Sclerosis Center, Columbus, Ohio, United States

REFERENCES:
- See also: The OSU MS Center — http://medicalcenter.osu.edu/patientcare/healthcare_services/multiple_sclerosis/